CLINICAL TRIAL: NCT04467463
Title: Comparing Two Peripheral Nerve Block Techniques for Perioperative Analgesia During Cleft Palate Surgery in Pediatric Patients: Randomized Controlled Trial
Brief Title: Peripheral Nerve Block Techniques During Cleft Palate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Elsonbaty, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: N-98-2019
Record Dates: First submitted 2020-07-04; First posted 2020-07-13 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-06

CONDITIONS: Postoperative Pain
Keywords: Suprazygomatic; Maxillary; Palatine; Cleft Palate
MeSH Terms: conditions — Pain, Postoperative; Cleft Palate | interventions — Levobupivacaine

STUDY DESIGN:
Intervention Model Description: The two study groups were:
  * Group GPN, 20 patients received bilateral greater palatine nerve block.
  * Group SMN, 20 patients received bilateral suprazygomatic maxillary nerve block.
Who Masked: Care Provider
Masking Description: masking from the aim of the study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GPN (Experimental): administrated bilateral greater palatine nerve block using levobupivacaine 0.25%
  Interventions: Procedure: peripheral nerve block by 0.25% levobupivacaine
- SMN (Experimental): administrated bilateral suprazygomatic nerve block using levobupivacaine 0.25%.
  Interventions: Procedure: peripheral nerve block by 0.25% levobupivacaine

INTERVENTIONS:
Procedure: peripheral nerve block by 0.25% levobupivacaine — SUBMANDIBULAR nerve block will be performed using a 25G 90 mm beveled needle . the entry point of the needle will be situated at the angle formed by the superior edge of the zygomatic arch below and the posterior orbital rim forward .The needle will be inserted perpendicular to the skin and advanced approximately 20 mm depth to reach the greater wing of the sphenoid deep to the pterygopalatine fossa. Injection of 1ml of 0.25% levobupivacaine will be done over 20 seconds afterensuring negative blood aspiration .greater Palatine Nerve will be blocked bilaterally as it leaves on palatal side through the foramen on the opposite direction of the anterior part of the 3rd molar orthe posterior part of the 2nd molar tooth.

SUMMARY:
Regional blocks are commonly used in pediatric anesthesia to achieve adequate postoperative analgesia. Suprazygomatic Maxillary nerve block (SMN) and Greater Palatine nerve block (GPN) are regional blocks described for use during cleft palate (CP) repair surgery.The aim of this study was to compare the analgesic effect as well as the incidence of complications associated with the use of bilateral GPN and bilateral SMN blocks in children undergoing palatoplasty surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III scheduled to undergo palatoplasty

Exclusion Criteria:

* bleeding disorders,
* skin lesions or wounds at site of proposed needle insertion,
* congenital heart disease,
* respiratory or
* cardiovascular disorders,
* children scheduled for combined procedures like palatoplasty with cheiloplasty or submucosal alveolar bone grafting,
* known hypersensitivity to local anesthetics or opioids and
* lack of parental consent.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
postoperative pain score | the first 12 postoperative hours
  Pain assessment was done immediately postoperative using Objective behavioral pain score

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Cairo University hospitals, Cairo, Manial
  - anesthesia department at Cairo University, Cairo

IPD SHARING:
Plan to Share IPD: No
not to share

REFERENCES:
- [Background] Pain terms: a list with definitions and notes on usage. Recommended by the IASP Subcommittee on Taxonomy. Pain. 1979 Jun;6(3):249. No abstract available. PMID 460932
- [Background] Lee SJ, Ralston HJ, Drey EA, Partridge JC, Rosen MA. Fetal pain: a systematic multidisciplinary review of the evidence. JAMA. 2005 Aug 24;294(8):947-54. doi: 10.1001/jama.294.8.947. PMID 16118385
- [Background] 3. Tremlett M. Anaesthesia for cleft lip and palate surgery. Curr Anaesth Crit Care. 2004;15:309-16.
- [Background] Diewert VM. Development of human craniofacial morphology during the late embryonic and early fetal periods. Am J Orthod. 1985 Jul;88(1):64-76. doi: 10.1016/0002-9416(85)90107-1. PMID 3860013